CLINICAL TRIAL: NCT07072000
Title: Shrinking the Anterior Border of CTV2 for Nasopharyngeal Carcinoma to Reduce the Radiation of Nasal Cavity : an Open-label, Non-inferiority, Multicenter, Randomized Phase III Trial
Brief Title: Shrinking the Anterior Border of CTV2 for Nasopharyngeal Carcinoma to Reduce the Radiation of Nasal Cavity
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hai-Qiang Mai,MD,PhD (Other)
Collaborators: First People's Hospital of Foshan (Other); Affiliated Hospital of Guangdong Medical University (Other); The Wuzhou Red Cross Hospital (Unknown); The Fourth Affiliated Hospital of Guangxi Medical University (Unknown); Zhongshan City People 's Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Hai-Qiang Mai,MD,PhD, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-FXY-483
Record Dates: First submitted 2025-07-16; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Nasopharyngeal Cancinoma (NPC)
Keywords: nasopharyngeal carcinoma; radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced delineation arm (Experimental)
  Interventions: Radiation: reduced CTV delineation
- Standard delineation arm (Active Comparator)
  Interventions: Radiation: standard CTV delineation

INTERVENTIONS:
Radiation: standard CTV delineation — The anterior border of CTV2 is delineated at the posterior 1/3 of the nasal cavity.
  Arms: Standard delineation arm
Radiation: reduced CTV delineation — The anterior border of CTV2 is defined as 5 mm anterior to the posterior nasal cavity anteriorly from the choanae.
  Arms: Reduced delineation arm

SUMMARY:
This is a an open-label, non-inferiority, multicenter, randomized phase III trial aimed to explore the efficacy and safety of shrinking the anterior border of CTV2 in nasopharyngeal carcinoma patients without tumor invasion into the posterior nasal aperture.

DETAILED DESCRIPTION:
This is a an open-label, non-inferiority, multicenter, randomized phase III trial aimed to explore the efficacy and safety of shrinking the anterior border of CTV2 in nasopharyngeal carcinoma patients without tumor invasion into the posterior nasal aperture. The enrolled patients will be 1:1 randomly assigned to receive reduced CTV delineation radiotherapy (anterior border of CTV2 defined as 5 mm anterior to the choanae), or standard CTV delineation radiotherapy (anterior border of CTV2 defined as the posterior 1/3 of the nasal cavity).

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed, histologically confirmed non-keratinizing carcinoma (WHO classification).
2. Stage I-III disease (AJCC 9th edition).
3. Tumor extends to nasal cavity (including nasal septum).
4. No distant metastasis (M0).
5. Age 18-70 years.
6. Male or non-pregnant female.
7. Scheduled for radiotherapy.
8. ECOG performance status 0-1 .
9. Adequate bone marrow function: white blood cells >4×10⁹/L, hemoglobin >90 g/L, platelets >100×10⁹/L.
10. Normal hepatic/renal function: total bilirubin ≤1.5×ULN, AST/ALT ≤2.5×ULN, alkaline phosphatase ≤2.5×ULN, creatinine clearance ≥60 mL/min.
11. Written informed consent obtained.

Exclusion Criteria:

1. Keratinizing squamous cell carcinoma (WHO Type I) or basaloid squamous cell carcinoma.
2. Age <18 or >70 years.
3. Recurrent disease or distant metastasis.
4. No tumor extension into the nasal cavity (including the nasal septum).
5. Prior malignancy (except adequately treated basal/squamous cell skin cancer or cervical carcinoma in situ).
6. Pregnancy/lactation (premenopausal women require pregnancy test; effective contraception mandated).
7. Prior radiotherapy (except non-melanoma skin cancer with lesions outside current portals).
8. Preoperative chemotherapy or surgical resection of primary/neck lesions (excluding diagnostic procedures).
9. Severe coexisting illness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2030-07-31 (Estimated); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
Local relapse-free survival | 3 year
  The time from randomization to documented local relapse or death from any cause.

SECONDARY OUTCOMES:
Overall survival | 3 year
  The time from randomization to death from any cause or censored at the date of the last follow-up.
Progression-free survival | 3 year
  The time from randomization to any documented local or regional relapse, distant metastasis, or death from any cause, whichever occur first.
Distant metastasis-free survival | 3 year
  The time from randomization to distant metastasis or death from any cause.
Regional relapse-free survival | 3 year
  The time from randomization to documented regional relapse or death from any cause.
Incidence rate of adverse events (AEs) | 2 year
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events(acute toxicity) as assessed by CTCAE v5.0.Numbers of patients of late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme.
Change of quality of life | 1 year
  Quality of life scores were assessed for each scale by using the 22-item Sino-Nasal Outcome Test (SNOT-22) before radiotherapy, at the end of radiotherapy, and at the 3, 6, 12 month after radiotherapy.

OTHER OUTCOMES:
Incidence of olfactory dysfunction | 1 year
  Olfactory function was assessed using the Visual Analogue Scale (VAS) before radiotherapy, at the end of radiotherapy, and at 3, 6, 12 month after radiotherapy.
Incidence of acquired nasal cavity stenosis and atresia | 1 year
  Acquired nasal cavity stenosis and atresia was assessed by electronic nasopharyngoscopy before radiotherapy, at the end of radiotherapy, and at 3, 6, and 12 months after radiotherapy.
Incidence of radiation-induced sinusitis | 1 year
  Radiation-induced sinusitis was assessed by head and neck enhanced magnetic resonance imaging (MRI) before radiotherapy, at the end of radiotherapy, and at 3, 6, and 12 months after radiotherapy.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - First People's Hospital of Foshan, Foshan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhangjiang, Guangdong
  - The Fourth Affiliated Hospital of Guangxi Medical University, Liuchow, Guangxi
  - Wuzhou Red Cross Hospital, Wuzhou, Guangxi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mao YP, Wang SX, Gao TS, Zhang N, Liang XY, Xie FY, Zhang Y, Zhou GQ, Guo R, Luo WJ, Li YJ, Liang SQ, Lin L, Li WF, Liu X, Xu C, Chen YP, Lv JW, Huang SH, Liu LZ, Li JB, Tang LL, Chen L, Sun Y, Ma J. Medial retropharyngeal nodal region sparing radiotherapy versus standard radiotherapy in patients with nasopharyngeal carcinoma: open label, non-inferiority, multicentre, randomised, phase 3 trial. BMJ. 2023 Feb 6;380:e072133. doi: 10.1136/bmj-2022-072133. PMID 36746459
- [Background] Sanford NN, Lau J, Lam MB, Juliano AF, Adams JA, Goldberg SI, Lu HM, Lu YC, Liebsch NJ, Curtin HD, Chan AW. Individualization of Clinical Target Volume Delineation Based on Stepwise Spread of Nasopharyngeal Carcinoma: Outcome of More Than a Decade of Clinical Experience. Int J Radiat Oncol Biol Phys. 2019 Mar 1;103(3):654-668. doi: 10.1016/j.ijrobp.2018.10.006. Epub 2018 Oct 15. PMID 30712708
- [Background] Lin SJ, Guo QJ, Liu Q, Ng WT, Ahn YC, AlHussain H, Chan AW, Chow J, Chua MLK, Corry J, Han F, Gregoire V, Harrington KJ, Hu CS, Jensen K, Langendijk JA, Le QT, Lee NY, Lee V, Lin JC, Ma J, Mendenhall WM, O'Sullivan B, Ozyar E, Rosenthal DI, Tao YG, Wang RS, Wee J, Xu ZY, Yi JL, Yom SS, Fan DM, Mai HQ, Pan JJ, Lee AWM. International Consensus Guideline on Delineation of the Clinical Target Volumes at Different Dose Levels for Nasopharyngeal Carcinoma (2024 Version). Int J Radiat Oncol Biol Phys. 2025 Oct 1;123(2):415-431. doi: 10.1016/j.ijrobp.2025.05.019. Epub 2025 May 24. PMID 40419028
- [Background] Lee NY, Zhang Q, Pfister DG, Kim J, Garden AS, Mechalakos J, Hu K, Le QT, Colevas AD, Glisson BS, Chan AT, Ang KK. Addition of bevacizumab to standard chemoradiation for locoregionally advanced nasopharyngeal carcinoma (RTOG 0615): a phase 2 multi-institutional trial. Lancet Oncol. 2012 Feb;13(2):172-80. doi: 10.1016/S1470-2045(11)70303-5. Epub 2011 Dec 15. PMID 22178121
- [Background] Liang SB, Sun Y, Liu LZ, Chen Y, Chen L, Mao YP, Tang LL, Tian L, Lin AH, Liu MZ, Li L, Ma J. Extension of local disease in nasopharyngeal carcinoma detected by magnetic resonance imaging: improvement of clinical target volume delineation. Int J Radiat Oncol Biol Phys. 2009 Nov 1;75(3):742-50. doi: 10.1016/j.ijrobp.2008.11.053. Epub 2009 Feb 27. PMID 19251378